CLINICAL TRIAL: NCT01527448
Title: An Open Label Dose Titration Study of Quetiapine XR in the Treatment of Postpartum Depression in Nonlactating Women Diagnosed With Bipolar Disorder (BD), Type II.
Brief Title: Quetiapine in the Treatment of Postpartum Depression (PPD) in Bipolar Disorder (BD), Type II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BC Women's Hospital & Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Shaila Misri, Principal Investigator, BC Women's Hospital & Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00032
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Postpartum Depression
Keywords: postpartum; postpartum depression; PPD; quetiapine XR; quetiapine; seroquel; bipolar; bipolar disorder; bipolar disorder, type II
MeSH Terms: conditions — Depression, Postpartum; Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atypical antipsychotic treatment (Experimental): Quetiapine XR is given to postpartum women diagnosed with bipolar disorder II. Starting dose is 50mg, maximum dose is 300mg/day.
  Interventions: Drug: Quetiapine XR (seroquel)

INTERVENTIONS:
Drug: Quetiapine XR (seroquel) — During the study period, subjects will be receiving a treatment with Quetiapine XR. The starting dose of quetiapine that subjects will receive is 50mg. The response to the treatment of quetiapine will determine whether the study doctor will increase the dosage of the subject's quetiapine. If the study doctor increases the quetiapine during the study, the maximum dosage allowable during the study is 300mg.
  Other Names: Seroquel XR

SUMMARY:
This is a 9-week single-centre, open-label, dose-escalating study evaluating the efficacy and safety of Quetiapine XR given as monotherapy in the treatment of non-lactating, post-partum women diagnosed with Bipolar II Disorder. Subjects will need to visit the study doctor up to 8 times over a period of 9 weeks.

During the study period, subjects will be receiving a treatment with Quetiapine XR. The starting dose of quetiapine that subjects will receive is 50mg. The response to the treatment of quetiapine will determine whether the study doctor will increase the dosage of the subject's quetiapine. If the study doctor increases the quetiapine during the study, the maximum dosage allowable during the study is 300mg.

DETAILED DESCRIPTION:
This study will help clinicians increase their awareness of the existence of Bipolar II Disorder in the perinatal population and provide guidance in terms of appropriate treatment. Since this diagnosis in the postpartum population is done by elimination, this study will provide evidence of the merits of identifying and treating this order on time. When selective serotonin reuptake inhibitors (SSRIs) fail for symptom relief in women diagnosed with unipolar depression, postpartum onset, clinicians tend to either augment or combine a variety of psychotropic medications for treatment response. It is probably likely that these patients are Bipolar II Disorder who continue to cycle through the treatment. Adding an atypical antipsychotic is often an afterthought. Therefore, the unique aspects of treating this specific population right at the outset when a diagnosis of mood disorders is made is optimal. Clinicians not only need to actively consider bipolar type II in their differential diagnosis, but also to initiate treatment as soon as possible to relieve further suffering. This study will help diagnose postpartum Bipolar II Disorder and test the unique action of quetiapine with its mood stabilizing and antidepressant properties.

Hypothesis:

Quetiapine XR will be effective in the treatment of postpartum depression in women with Bipolar II Disorder.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent;
* women, 19 - 40 years;
* meets Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria of Bipolar II Disorder (confirmed by Mini International Neuropsychiatric Interview (MINI));
* Hamilton Depression Rating Scale (HAM-D) (17-item) total score of > 22 and HAM-D item 1 (depressed mood) score of >2 at Visit 1 (enrolment) & Visit 2;
* negative serum pregnancy test at enrolment, use reliable method of birth control (i.e. barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal ligation) during study;
* understand and comply with requirements of study
* outpatient status at enrolment.

Exclusion Criteria:

* DSM-IV Axis I disorder other than Bipolar II Disorder within 6 months of enrolment;
* diagnosis of DSM-IV Axis II disorder which has a major impact on the patient's current psychiatric status;
* substance or alcohol abuse or dependence within 6 months prior to enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined in DSM-IV criteria;
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment;
* use of drugs that induce or inhibit the hepatic metabolizing cytochrome P450 3A4 enzymes within 2 weeks prior to Visit 2;
* pregnancy or lactation;
* evidence of clinically relevant disease, e.g., renal or hepatic impairment, significant coronary artery disease, cerebrovascular disease, viral hepatitis B or C, acquired immunodeficiency syndrome (AIDS);
* clinical finding that is unstable or inadequately treated, (e.g., hypertension, poorly controlled diabetes, unstable angina) or that would be negatively affected by the study medication or affect the study medication;
* medical conditions that would affect absorption, distribution, metabolism, or excretion of study medication (e.g., malabsorption syndrome, liver disease);
* current diagnosis of cancer (except basal or squamous cell skin carcinoma) unless in remission for at least 5 years;
* current or past diagnosis of stroke or Transient Ischemic Attacks (TIA);
* history of seizure disorder, except febrile convulsions;
* receipt of electroconvulsive therapy (ECT) within 90 days prior to Visit 2;
* use of antipsychotic, mood stabilizer, or antidepressant drugs within 7 days before Visit 2, or use of fluoxetine within 28 days before Visit 2, or use of monoamine oxidase inhibitors (MAOIs), anxiolytic or hypnotics within 14 days before Visit 2 (with the exception of those allowed with restriction per protocol), or use of a depot antipsychotic injection within 2 dosing interval before Visit 2;
* subjects who will require psychotherapy (other than supportive psychotherapy) during the study period, unless psychotherapy has been ongoing for a minimum of 3 months prior to Visit 2;
* subjects who pose a current serious suicidal or homicidal risk, have a HAM-D item 3 score of 3 or greater, or have made a suicide attempt within the past 6 months;
* a patient with Diabetes Mellitus (DM) fulfilling specific criteria as judged by the investigator that would make her unable to participate;
* clinically significant deviation from the reference range in clinical laboratory test results as judged by the investigator;
* an absolute neutrophil count (ANC) of <1.5 x 109 per liter;
* a thyroid-stimulating hormone (TSH) concentration more than 10% above the upper limit of the normal range of the laboratory used for sample analysis at enrolment, whether or not the patient is being treated for hypothyroidism;
* liver function tests aspartate aminotransferase (AST) or alanine aminotransferase (ALT) three times the upper normal limit;
* Electrocardiogram (ECG) results considered being clinically significant based on assessment by a centrally located experienced cardiologist interpreting the ECG;
* use of quetiapine in doses greater than 25mg/day for insomnia within 7 days before Visit 2;
* known history of intolerance or hypersensitivity to quetiapine;
* known lack of response to quetiapine in the treatment of depression in a dosage of at least 50 mg per day for 4 weeks (at any time before study start);
* treatment with quetiapine with a dosage of at least 50 mg/day at Visit 1 (enrolment);
* contraindications as detailed in the country-specific prescribing information for quetiapine;
* involvement in the planning and conduct of the study;
* previous enrolment in any AstraZeneca-sponsored study with quetiapine;
* participation in another clinical study or compassionate use programme within 4 weeks of Visit 2 or longer in accordance with local requirements.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy assessment will be total score on the Montgomery-Asberg Depression Rating Scale (MADRS). | The primary variable is the change from Week 0 to Week 8 in the MADRS score

SECONDARY OUTCOMES:
To evaluate if Quetiapine XR improves the health relate quality of life of postpartum depression in non-lactating women with Bipolar II Disorder | Change from Week 0 to Week 8 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) total score. Change from Week 0 to Week 8 in Q-LES-Q Item 16 (Overall quality of life) score.
To evaluate if Quetiapine XR improves satisfaction with medication in postpartum depression in non-lactating women with Bipolar II Disorder. | Change from Week 0 to Week 8 in Q-LES-Q Item 15 (Satisfaction with medication) score.
To evaluate if Quetiapine XR improves sleep quality in postpartum depression in non-lactating women with Bipolar II Disorder. | Change from Week 0 to Week 8 in Pittsburgh Sleep Quality Index (PSQI) global score.

CONTACTS AND LOCATIONS:
Overall Officials: Shaila Misri, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada